CLINICAL TRIAL: NCT07353983
Title: Pharmacokinetic Evaluation of Anrikefon Injection in the Geriatric Population With the Management of Acute Pain Following Abdominal Laparoscopy
Acronym: PAGAP1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025 1539
Record Dates: First submitted 2025-11-19; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The age group of 65 to 74 years old (Experimental)
  Interventions: Drug: Inject Anrikefon Injection
- Age group ≥75 years old (Experimental)
  Interventions: Drug: Inject Anrikefon Injection

INTERVENTIONS:
Drug: Inject Anrikefon Injection — After the end of the operation ( the end of the last needle suture ), the researchers need to give the subjects 1.0μg / kg of Anrikefon Injection for the first time as soon as possible ( within 15 minutes ) ( 1ml of Anrikefon Injection stock solution was diluted to 10ml, and then the dose was calculated according to the body weight, and the corresponding volume was extracted, and the injection was completed in about 2 minutes ).

SUMMARY:
This study used a single-center, single-arm, pharmacokinetic ( PK ) study design. Thirty subjects who met the inclusion criteria were stratified according to age, including 15 in each age group of 65-74 years old and ≥ 75 years old. The patients were treated with a unified anesthesia method during abdominal endoscopic surgery. Anrecofin injection 1.0 μg / kg was injected for the first time within 15 min, and then once again at 8 h and 16 h. And received 6 pain assessments, 1 satisfaction score and 1 telephone follow-up. In this study, 10 blood samples were collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years, gender unrestricted;
* American Society of Anesthesiologists (ASA) classification I-III;
* 18 kg/m2 ≤ BMI < 30 kg/m2;
* Undergoing elective general anesthesia for laparoscopic surgery and expected to experience mild to moderate postoperative pain;
* Agree to participate in this trial and voluntarily sign the informed consent form.

Exclusion Criteria:

* There is a history or evidence of any of the following diseases before screening:1) History of cardiovascular diseases: Uncontrolled hypertension (systolic blood pressure ≥160 MMHG and/or diastolic blood pressure ≥90mmHg), as well as a history of cardiovascular diseases evaluated by the researcher as unsuitable for participation in the study, such as severe arrhythmia, heart failure, acute myocardial ischemia, unstable angina pectoris, myocardial infarction, II-III degree atrioventricular block, etc.2) Respiratory system history: Severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe airway stenosis, and other respiratory system histories assessed by the researcher as unsuitable for participation in the study;3) History of neurological and mental system diseases: Craniocerebral injury, intracranial hypertension, schizophrenia, mania, cognitive dysfunction, etc., evaluated by the researcher as unsuitable for participation in the study;4) History of digestive system diseases: Suffering from intestinal obstruction or other digestive system diseases that the researcher deems may cause nausea and vomiting;5) Accompanied by a clear history of chronic dizziness, or clearly diagnosed vestibular dysfunction other than motion sickness (including but not limited to: peripheral vestibular syndrome, central vestibular syndrome, etc.);6) Tumor patients who have received chemotherapy and/or radiotherapy within 4 weeks prior to being informed.
* It is expected that tracheal intubation will continue after the operation or a nasal or oral gastric tube will need to be inserted.
* Known to be allergic or contraindicated to opioid drugs and other anesthetics and antiemetic drugs that may be used during the trial;
* Within 3 months prior to screening, there is a history of drug abuse, or continuous use of opioid analgesics for more than 10 days for any reason;
* Abnormal liver and kidney functions:1) Prothrombin time (PT) is prolonged by more than 3 seconds beyond the upper limit of the normal value;2) Alanine aminotransferase and/or aspartate aminotransferase > 2×ULN;3) Total bilirubin > 1.5×ULN;4) Glomerular filtration rate (eGFR) < 60 mL/min.
* Have participated in any clinical researchers within the three months prior to the screening;
* Pregnant and lactating women who have plans to become pregnant during the study period or within 3 months after the study ends;
* Subjects who the researchers consider to have any other factors that make them unsuitable for participating in this clinical study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-22 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood concentration | The blood collection time points were Minute 0, Minute 2, Minute 5, Minute 10, Minute 30, Hour 1, Hour 2, Hour 4, Hour 8, Hour 12 after the 3rd intravenous injection.
  Determine the blood concentration of the Anrikefon using liquid chromatography technology.

IPD SHARING:
Plan to Share IPD: Undecided